CLINICAL TRIAL: NCT03836846
Title: Social Media Use in Adolescents Admitted to a Psychiatric Unit
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not initiated because it was not approved by KPSC IRB.
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 029021
Record Dates: First submitted 2019-02-08; First posted 2019-02-11 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Depression; Social Media; Adolescent Behavior
MeSH Terms: conditions — Depression; Adolescent Behavior | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment As Usual (Placebo Comparator): Standard of care as usual with follow-up at 1-, 3-, and 6-months
  Interventions: Behavioral: Treatment as usual
- Intervention with CBT Mobile App (Active Comparator): Treatment as usual with additional treatment using cognitive behavioral therapy (CBT) mobile apps (ie What's Up?)
  Interventions: Behavioral: CBT Mobile App

INTERVENTIONS:
Behavioral: CBT Mobile App — TAU and the additional treatment of a Mental Health App (What's Up?). This app will be used to guide adolescents through cognitive behavioral therapy and acceptance commitment therapy techniques, as well as to assist in developing coping mechanisms to prevent readmission.
  Arms: Intervention with CBT Mobile App
Behavioral: Treatment as usual — TAU as per standard of care
  Arms: Treatment As Usual

SUMMARY:
We will investigate the association between social media use and depression in adolescents admitted to a psychiatric unit and continue to follow their progress after discharge in outpatient clinic services. We expect improvement in their depressive symptoms by modifying social media use and adding a mental health app to further encourage the positive effects of social media.

ELIGIBILITY:
Inclusion Criteria:

* Participants admitted to inpatient psychiatric unit
* Kaiser insured participants between 13-17 years of age with parental consent
* positive for social media use
* English speaking

Exclusion Criteria:

* pregnant
* non English speaking

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Comparing depression scale,PHQ9-A (Patient Health Questionnaire, Adolescent Version), with social media use | 1 month
  Compare presence and severity of depressive symptoms in treatment as usual (TAU) group with TAU and the mobile app intervention group. The presence and severity of depression will be determined using the PHQ9-A (Patient Health Questionnaire, adolescent version), a 9-question depression scale that is based on the DSM-IV diagnostic criteria of depression and modified for teens to further inquire about other aspects of depression such as dysthymia, suicide risk, and other mental illnesses. The PHQ-9A scores each of the DSM-IV criteria as "0" (not at all) to "3" (nearly every day). Total depression severity score ranges of 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.
Comparing depression scale,PHQ9-A (Patient Health Questionnaire, Adolescent Version), with social media use | 3 months
  Compare presence and severity of depressive symptoms in treatment as usual (TAU) group with TAU and the mobile app intervention group. The presence and severity of depression will be determined using the PHQ9-A (Patient Health Questionnaire, adolescent version), a 9-question depression scale that is based on the DSM-IV diagnostic criteria of depression and modified for teens to further inquire about other aspects of depression such as dysthymia, suicide risk, and other mental illnesses. The PHQ-9A scores each of the DSM-IV criteria as "0" (not at all) to "3" (nearly every day). Total depression severity score ranges of 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.
Comparing depression scale,PHQ9-A (Patient Health Questionnaire, Adolescent Version), with social media use | 6 months
  Compare presence and severity of depressive symptoms in treatment as usual (TAU) group with TAU and the mobile app intervention group. The presence and severity of depression will be determined using the PHQ9-A (Patient Health Questionnaire, adolescent version), a 9-question depression scale that is based on the DSM-IV diagnostic criteria of depression and modified for teens to further inquire about other aspects of depression such as dysthymia, suicide risk, and other mental illnesses. The PHQ-9A scores each of the DSM-IV criteria as "0" (not at all) to "3" (nearly every day). Total depression severity score ranges of 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Canyon Ridge Hospital, Chino, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
All data will be collected by trained study personnel, and each study participant will be assigned a unique study number. Data will be de-identified after collection and hard copies of data will be stored in a locked cabinet in the investigator's office. We are considering options to share de-identified data.

REFERENCES:
- [Background] Pantic I. Online social networking and mental health. Cyberpsychol Behav Soc Netw. 2014 Oct;17(10):652-7. doi: 10.1089/cyber.2014.0070. Epub 2014 Sep 5. PMID 25192305
- [Background] Luxton DD, June JD, Fairall JM. Social media and suicide: a public health perspective. Am J Public Health. 2012 May;102 Suppl 2(Suppl 2):S195-200. doi: 10.2105/AJPH.2011.300608. Epub 2012 Mar 8. PMID 22401525
- [Background] Banos RM, Etchemendy E, Mira A, Riva G, Gaggioli A, Botella C. Online Positive Interventions to Promote Well-being and Resilience in the Adolescent Population: A Narrative Review. Front Psychiatry. 2017 Jan 30;8:10. doi: 10.3389/fpsyt.2017.00010. eCollection 2017. PMID 28194117
- See also: Teens, Social Media & Technology 2018 — http://www.pewinternet.org/2018/05/31/teens-social-media-technology-2018/
- See also: Social media and young people's mental health and wellbeing — https://www.scie-socialcareonline.org.uk/statusofmind-social-media-and-young-peoples-mental-health-and-wellbeing/r/a110f00000NeITGAA3